CLINICAL TRIAL: NCT03751592
Title: A Single Arm, Open-label, Multicenter, Phase Ib/IIa Studies of Chlorogenic Acid for Injection for Safety and Efficacy of Advanced Lung Cancer Patients
Brief Title: Phase Ib/IIa Studies of Chlorogenic Acid for Injection for Safety and Efficacy of Advanced Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan J.Z. Bio-chemical Science and Technology Development Co., Ltd (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYS-LC-01
Record Dates: First submitted 2018-11-19; First posted 2018-11-23 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-09

CONDITIONS: Advanced Lung Cancer
MeSH Terms: interventions — Chlorogenic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chlorogenic acid, Treatment, powder (Experimental): Chlorogenic acid for injection(30mg/bottle) is white or off-white freeze-dried lump or powder,it can be easily dissolved in water, which solubility is 20%.
  Interventions: Drug: Chlorogenic acid

INTERVENTIONS:
Drug: Chlorogenic acid — Chlorogenic acid for injection is polyphenols, micromolecular and un-endogenous substance. It might play the role of cancer treatment via balancing tumor micro-environmental immune status according to the stability and rationality of immunodeficiency and endogenous immune material expression around the tumor. Chlorogenic acid for injection is made from chlorogenic acid (purity≥98%) which is extracted from folium cortex eucommiae.Chlorogenic acid and its preparations have not been reported as chemical drug and marketed around the world.

SUMMARY:
This Ib / IIa clinical trial program focuses on the small cell lung cancer (SCLC), Squamous non-small cell lung cancer (NSCLC) and adeniform NSCLC in order to start a better development on the broad-spectrum value of chlorogenic acid： Determine the Disease control rate（DCR）of phase Ib/IIa of Chlorogenic acid for injection in the advanced Lung Cancer Patients.

DETAILED DESCRIPTION:
1. Determine the Disease control rate（DCR）of Chlorogenic acid for injection in the advanced Lung Cancer Patients;
2. Determine the Overall Survival（OS）of Chlorogenic acid for injection in the advanced Lung Cancer Patients;
3. Determine the Objective response rate（ORR）of Chlorogenic acid for injection in the advanced Lung Cancer Patients;
4. Determine the Progression Free Survival（PFS）of Chlorogenic acid for injection in the advanced Lung Cancer Patients;
5. Determine Eastern Cooperative Oncology Group（ECOG）.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18;
2. Recurrent small cell lung cancer (SCLC), Squamous non-small cell lung cancer (NSCLC) and adeniform NSCLC;
3. Estimated lifetime ≥ 3 months；
4. Patients who have sufficient baseline organ function and whose laboratory data can meet the following criteria at the enrollment:1)PLT count≥80×10~9/L； 2)NEUT# count≥1.5×10~9/L ；3)HGB count≥90g/L；4)Total bilirubin <=1.5 times of ULN；5)ALT/AST ≤2.5 times of ULN；
5. Female patients with negative pregnant test, and male/female patients of reproductive age without pregnancy planning in the next 12 months;
6. Volunteered for the phase 1 trial and sign the informed consent without protest.

Exclusion Criteria:

1. Patients who suffer from other serious complication, such as uncontrollable infection, myocardial infarction within the past 6 months at the enrollment , uncontrollable hypertension ,thromboembolism and etc.;
2. Patients with brain metastases;
3. Patients with bone metastases;
4. Patients who have primary immunodeficiency;
5. Organ transplanters recipients;
6. Patients who have received the therapy of chemotherapy within 4 weeks or radical radiotherapy with in 6 weeks before enrollment;
7. Pregnant or breast-feeding women, or patients(male and female) who have pregnancy plan;
8. Patients who had received a therapy of another investigational drug within 1 month；
9. Known active hepatitis B/hepatitis C, positive HIV/ syphilis antibody;
10. Patients who have received therapy of major surgery within 6 weeks or biopsy surgery within 2 weeks before enrollment;
11. Patient who need long term treatment of cortical hormone or other immunosuppressive drugs such as visceral organ transplanters；
12. Patients who have used nitrosoureas drug or mitomycin within 6 weeks or tyrosine kinase inhibitor within 2 weeks before enrollment;
13. Patients who or have received radical radiotherapy within 6 weeks or local palliative radiotherapy within 2 weeks before enrollment;
14. History of drug abuse；
15. Patients who was treated with Immunologic drugs in 3 months;
16. Other patients judged ineligible for enrollment in the study by the investigator (sub-investigator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2018-07-17 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
disease control rate（DCR) | Within the first 10 weeks after the first dose of chlorogenic acid for injection

SECONDARY OUTCOMES:
objective response rate (ORR) | Within the first 10 weeks after the first dose of chlorogenic acid for injection
progress free survival(PFS) | Within the first 10 weeks after the first dose of chlorogenic acid for injection
Overall Survival（OS） | Within the first 10 weeks after the first dose of chlorogenic acid for injection
Eastern Cooperative Oncology Group （ECOG） score standard | Within the first 10 weeks after the first dose of chlorogenic acid for injection

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Dr, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No